CLINICAL TRIAL: NCT03797183
Title: The Associations Between EIT and Clinical Measures During Standard of Care Procedures in Patients With Respiratory Disease: A Preliminary Study
Brief Title: Genesis Electrical Impedance Tomography (EIT): A Preliminary Study
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 18-1843
Record Dates: First submitted 2018-12-28; First posted 2019-01-09 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Premature Infant; Chronic Respiratory Disease; Neuromuscular Diseases; Healthy; Bronchopulmonary Dysplasia; Pulmonary Vein Stenoses
MeSH Terms: conditions — Premature Birth; Neuromuscular Diseases; Bronchopulmonary Dysplasia; Stenosis, Pulmonary Vein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Premature Infants: Premature infants >1 month of age currently hospitalized with bronchopulmonary dysplasia (BPD) without acute respiratory infection
- Chronic Respiratory Disease: Participants ages >1 month-21 years with chronic respiratory disease due to underlying neuromuscular disease
- Neuromuscular Disease: Participants ages 21-40 years with confirmed neuromuscular disease with an echo completed within the preceding 12 months of study participation of Duchenne muscular dystrophy (DMD) or other diagnoses associated with mild cardiomyopathy
- Healthy Controls: Age and height matched healthy controls
- V/Q Scan validation: Adults or children who are having or have recently had a V/Q scan
- Premature Infants (Longitudinal Cohort): Premature infants ages 2 weeks to 1 year with diagnosed or suspected bronchopulmonary dysplasia
- Pulmonary Vein/Artery Stenosis: Children age 2 months to 18 years, who will be undergoing cardiac catheterization for pulmonary vein stenosis, pulmonary hypertension and/or pulmonary artery stenosis

SUMMARY:
The purpose of this study is to evaluate the Genesis Electrical Impedance Tomography (EIT) imaging system for use in pediatric respiratory disease populations including neuromuscular and bronchopulmonary dysplasia, as well as in age and height matched controls. The EIT does not use radiation, and is read through electrodes.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate EIT for use in pediatric respiratory disease populations including neuromuscular and bronchopulmonary dysplasia, as well as in age and height matched controls.

Researchers will use EIT to determine changes in regional ventilation with pulmonary interventions including airway clearance and invasive and noninvasive ventilation in a pediatric respiratory disease population.

ELIGIBILITY:
Inclusion Criteria:

* 2 weeks old - 40 years old
* Premature infants with current age >2 weeks with a confirmed diagnosis of BPD based on NIH criteria
* Or Chronic respiratory disease due to underlying neuromuscular disease
* Or confirmed neuromuscular disease with an echo completed within the preceding 12 months of study participation of DMD or other diagnoses associated with mild cardiomyopathy.
* have had a VQ scan
* will be undergoing cardiac catherization for for pulmonary vein stenosis, pulmonary hypertension and/or pulmonary artery stenosis
* Or healthy controls

Exclusion Criteria:

* <2 weeks of age
* Congenital diaphragmatic hernia
* Severe congenital heart disease
* Significant genetic abnoralities
* Anything that interferes with lead placement on the chest wall
* Unwilling/refusal to sign consent
* Pregnant or lactating
* Pacemaker of other surgical implant and spinal implant (causes noise in the data)
* Moderate to severe cardiomyopathy
* Patients with temporary cognitive disability due to illness

Ages: 14 Days to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: pediatric respiratory disease populations including neuromuscular and bronchopulmonary dysplasia, as well as in age and height matched controls. Populations who will be undergoing cardiac catheterization for pulmonary vein stenosis, pulmonary hypertension and/or pulmonary artery stenosis
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-05-03 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
EIT imaging maps that provide regional information regarding ventilation and perfusion of the lung. | 24 months
  These images will be analyzed both visually for qualitative abnormalities and through quantitative pixel analysis that can provide information regarding lung volume, blood volume, and changes in either based on respiratory cycle, cardiac cycle, or intervention. Areas of low ventilation (atelectasis and consolidation) will be identified.

SECONDARY OUTCOMES:
Regional conductivity changes due to ventilation | 24 months
  Describe regional ventilation in pediatric respiratory disease populations including neuromuscular weakness, skeletal/chest wall disorders, and chronic airway and parenchymal lung disease including bronchopulmonary dysplasia.
  This is a qualitative aim and will summarize EIT images pictorially. Pixel densities will be evaluated for normality and summarized as mean (SD) or median (interquartile range). EIT images will be qualitatively compared between cases and controls.
Waveform for a mesh element | 24 months
  Time-series waveform indicated by time in seconds compared to Recon signal (au).
Regional conductivity changes due to perfusion | 24 months
  This is a qualitative and quantitative aim. Results will qualitatively compare EIT images with CXR and CT scan images when available. Images will be displayed side by side and interpreted by both the clinician and the EIT study staff. Various summary measures of EIT outcomes will be calculated including pixel heterogeneity, summary changes over tidal breath and variation between tidal peaks. Pearson and Spearman correlation will be calculated between summary EIT outcomes and continuous primary clinical values. Linear and logistic regression will be used to estimate associations (with 95% CI) between EIT measures and clinical outcomes. Summary data will be presented in tables and figures using basic descriptive statistics stratified by study group.
Regional pulsatile perfusion imaging at the end of systole | 5 minutes
Power waveform (computed as the inner product of measured voltages and applied currents) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No